CLINICAL TRIAL: NCT06935721
Title: An Open-label, Single-dose, Three-period Phase 1 Study to Compare the Pharmacokinetics of Y-4 Tablets With Pregabalin Capsules and Riluzole Tablets in Healthy Subjects Under Fasted Condition
Brief Title: Pharmacokinetics of Y-4 Tablets With Pregabalin Capsules and Riluzole Tablets in Chinese Healthy Subject
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Beijing Tiantan Hospital (Other)
Collaborators: Neurodawn Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Yongjun Wang, Chief Physician, Beijing Tiantan Hospital
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: Y-4-LC-02
Record Dates: First submitted 2025-04-02; First posted 2025-04-20 (Actual); Last update posted 2025-04-20 (Actual); Status verified 2025-04

CONDITIONS: Healthy Male and Female Subjects
Keywords: phase I trial
MeSH Terms: interventions — Pregabalin; Riluzole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Y-4 tables (Experimental): Single oral administration in the state of fasting state
  Interventions: Drug: Y-4 tablet
- Pregabalin capsules (Experimental): Single oral administration in the state of fasting state
  Interventions: Drug: Pregabalin capsule
- Riluzole tablets (Experimental): Single oral administration in the state of fasting state
  Interventions: Drug: Riluzole tablet

INTERVENTIONS:
Drug: Y-4 tablet — Subjects will be admitted to research center in the afternoon of Day-1 prior to the dosing day and fasting for the next 10 hours overnight. In the morning of the following day (Day 1), subjects will be administered with one tablet of Y-4 , then subjects will be monitored and blood samples will be collected for the following 72 hours. Subjects will be discharged on Day 4.
  Arms: Y-4 tables
Drug: Pregabalin capsule — Subjects will be admitted to research center in the afternoon of Day 7 prior to the dosing day and fasting for the next 10 hours overnight. In the morning of the following day (Day 8), subjects will be administered with one pregabalin capsule , then subjects will be monitored and blood samples will be collected for the following 72 hours. Subjects will be discharged on Day 11.
  Arms: Pregabalin capsules
Drug: Riluzole tablet — Subjects will be admitted to research center in the afternoon of Day 14 prior to the dosing day and fasting for the next 10 hours overnight. In the morning of the following day (Day 15), subjects will be administered with one riluzole tablet, then subjects will be monitored and blood samples will be collected for the following 72 hours. Subjects will be discharged on Day 18 after safety evaluation.
  Arms: Riluzole tablets

SUMMARY:
Y-4 is a new fixed-dose combination drug product containing two active ingredients of pregabalin and riluzole.

The objective of the trial is to compare pharmacokinetic characteristics of Y-4 tablets with pregabalin capsules (Lyrica®) and riluzole tablets (Rilutek®) in Chinese healthy adult subjects after single oral administration under fasted condition.

DETAILED DESCRIPTION:
This study will be an open-label, single-dose, three-period study in healthy adult subjects. A total of 10 subjects (half men and half women) will be enrolled in this study to be administered with Y-4 tablets, pregabalin capsules and riluzole tablets at three periods with a 7-day washout.

Periods and corresponding treatments are planned as following:

Period 1: Y-4 tablet, one tablet, 112.5 mg/28.125 mg (pregabalin/riluzole) Period 2: pregabalin capsule, one capsule, 75 mg/capsule Period 3: riluzole tablet, one tablet, 50 mg/tablet

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adult male and female subjects, 18-45 years of age (including both ends).
2. Body weight ≥ 50 kg for male and ≥ 45 kg for female, body mass index (BMI) within the range of 19 - 28 kg/m2 (including both ends).
3. During the screening period, serum creatinine is within the normal range, or the standard creatinine clearance (CLcr) estimated by Cockcroft-Gault formula is ≥ 80 mL/min (for female subject, according to the calculation result × 0.85）.
4. Subjects who are able to understand and give their signed informed consent before any trial related procedures are performed.

Exclusion Criteria:

1. Subjects who are known to be allergic to pregabalin, riluzole or any excipients of Y-4 tablets (microcrystalline cellulose, Copovidone, croscarmellose sodium, colloidal silicon dioxide, magnesium stearate and Opadry amb Ⅱ), have allergic diseases or allergic constitution;
2. Subjects who have special requirements for diet and cannot follow the unified diet;
3. Physical examinations, vital signs, 12-lead electrocardiograms (ECG), chest X-ray (front position), laboratory tests (hematology, serum chemistry, coagulation test, urinalysis, etc.) and other screening tests found abnormalities that the researchers judged to be of clinical significance;
4. Subjects who have experienced angioedema in the past (such as swelling of the face, mouth (tongue, lips, and gums), and neck (pharynx and throat));
5. History of dizziness or vertigo with clinical significance, or disease of inner ear known to cause dizziness or vertigo;
6. QTcF > 450 msec at the screening stage;
7. Diagnosed with insomnia, anxiety disorder, depression, epilepsy, or other serious mental disorders, and principal investigator determines that the subject is not suitable to participate in this trial;
8. Presence or history of hepatic or renal disease or any other condition known to interfere with the absorption, distribution, metabolism or excretion of medicines;
9. Subjects who drink too much tea, coffee and/or caffeine-containing beverages (more than 8 cups, 1 cup = 250 mL) every day within 3 months prior to screening, or disagree that any caffeine-containing beverages are prohibited during the trial;
10. Subjects who have consume any diet (food or beverage) rich in grapefruit, pitaya, mango and cranberry within 14 days prior to screening;
11. Subjects have disease history or current disease that may affect the safety evaluation of the subject or the internal process of the study drug, including the central nervous system, cardiovascular system, digestive system, respiratory system, urinary system, hematological system, immunology, psychiatry, metabolic abnormalities, gastrointestinal surgery (excluding appendicitis surgery), etc. In particular, there is a history of dysphagia or any gastrointestinal disease affecting drug absorption (including frequent nausea or vomiting caused by any cause) and eye diseases;
12. Donation or loss of blood equal to or in excess of 400 mL, or blood transfusion within 3 months prior to screening; or donation or loss of blood equal to or in excess of 200 mL within 1 month prior to screening;
13. Subjects who have taken any drugs known to be strong inhibitors or inducers of cytochrome P450 enzymes within 2 months prior to screening (such as inducers - barbiturates, carbamazepine, phenytoin, glucocorticoids, omeprazole; inhibitors - serotonin reuptake inhibitors (SSRI) antidepressants, cimetidine, diltiazem, macrolides, nitroimidazoles, sedative hypnotics, verapamil, fluoroquinolones, antihistamines); or subjects who have taken any prescription drugs, over-the-counter drugs and Chinese herbal medicine other than the above drugs within 14 days prior to screening;
14. Subjects who have taken central nervous system (CNS) depressants including opioids (pethidine hydrochloride, morphine, dihydromorphine hydrochloride, fentanyl, tramadol, etc), benzodiazepines (diazepam, flurazepam, clonazepam, oxazepam, chlordiazepine and triazolam etc), antiepileptic drugs (carbamazepine, sodium valproate, phenobarbital drugs etc) within 2 months prior to screening;
15. Subject with sleep apnea, or subjects with severe sleep snoring and daytime drowsiness;
16. Subjects with suicidal thoughts and behavior;
17. Subject participated in any other clinical trials within 3 months prior to screening;
18. Current or former drug users, or positive urine screen for drugs of abuse at screening (screening items include: dimethylenedioxyamphetamine, methamphetamine, ketamine, morphine, tetrahydrocannabinoid acid, cocaine);
19. Alcoholics or regular drinkers within 3 months prior to screening, that is, those who drink more than 14 units of alcohol per week (1 unit = 360 mL of beer or 45 mL of alcohol with 40% alcohol content or 150 mL of wine), or whose alcohol breath test results are greater than 0.0 mg/100 mL, or who cannot abstain from alcohol during the trial;
20. Smokers or those who cannot comply with the prohibition of smoking during the trial, or positive for cotinine screening;
21. Subjects who is positive for hepatitis B surface antigen (HBsAg), hepatitis C virus (HCV) antibody, syphilis antibody or human immunodeficiency virus (HIV) antibody;
22. Male subjects (or their partners) or female subjects have baby plans during the whole trial period and within 3 months after the end of the trial, or subjects are unwilling to take one or more non-drug contraceptive measures (such as complete abstinence, condoms, ligation, etc.) during the trial period;
23. Female subjects who have unprotected intercourse within 14 days prior to screening, or pregnant or lactating women;
24. Subjects with poor compliance or other factors unsuitable for participation in this trial.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-03-28 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
adverse events | From the first day to the 25th± 1st day after the start of administration
  An AE is defined as any untoward medical event that occurs after receiving a drug or treatment or any deterioration of a disease or symptom that existed before receiving the investigational product or treatment (excluding the disease studied in this trial) in a subject or a clinical investigation subject, whether or not considered related to the investigational product or treatment. Therefore, an AE can be a discomfort sign (including an abnormal laboratory finding), symptom, or transient disease beyond any indication, whether or not related to the investigational product or treatment. The investigator will name each AE reported during the study by MedDRA PT and evaluate their severity using the criteria of "mild", "moderate" and "severe". The relevance evaluation is divided into 5 grades: 1-certainly related; 2- probably/likely related; 3-possibly related; 4-unlikely related; 5 not related.
Incidence of subject getting abnormal results of laboratory tests after treatment | From the first day to the 25th± 1st day after the start of administration
  Record changes from baseline to post-treatment, listing deviations from normal ranges post-treatment. Laboratory tests are composed of hematology, urinalysis, serum chemistry, coagulation test. Normal range is provided by the site.
Incidence of subject getting abnormal results of 12-lead ECG after treatment | From the first day to the 25th± 1st day after the start of administration
  Record changes from baseline to post-treatment, listing deviations from normal ranges post-treatment. 12-lead ECG will be analyzed by single RR Heart Rate, aggregate PR Interval, aggregate QRS Duration, aggregate RR Interval, aggregate QT Interval, aggregate QTC Interval. Normal range is provided by the site.
Incidence of subject getting abnormal results of vital signs after treatment. | From the first day to the 25th± 1st day after the start of administration
  Record changes from baseline to post-treatment, listing deviations from normal ranges post-treatment. Vital signs(body temperature, respiration, blood pressure, and pulse) will be assessed by according equipment.(electronic sphygmomanometer, thermometer).
Incidence of subject getting abnormal results of physical examinations after treatment. | From the first day to the 25th± 1st day after the start of administration
  Record changes from baseline to post-treatment, listing deviations from normal ranges post-treatment. Physical examinations will be conduct by the investigator through observation.
Incidence of subject getting abnormal results of blood oxygen saturation after treatment | From the first day to the 25th± 1st day after the start of administration
  Record changes of blood oxygen saturation from baseline to post-treatment, listing deviations from normal ranges post-treatment. Normal range is provided by the site
Incidence of subject getting abnormal results of C-SSSRS scale evaluation after treatment after treatment | From the first day to the 25th± 1st day after the start of administration
  Record changes of C-SSSRS scale evaluation from baseline to post-treatment

SECONDARY OUTCOMES:
Cmax | Up to 72 hours post-dose of each drug
  peak plasma concentration
AUC0-t | Up to 72 hours post-dose of each drug
  Area under the plasma concentration versus time curve from time 0 to the time of the last quantifiable concentration
AUC0-∞ | Up to 72 hours post-dose of each drug
  Area under the plasma concentration-time curve from time 0 to infinity (extrapolated)
Tmax | Up to 72 hours post-dose of each drug
  Time to reach maximum observed plasma concentration after single dose
t1/2 | Up to 72 hours post-dose of each drug
  Terminal elimination half-life after single dose
λz | Up to 72 hours post-dose of each drug
  Terminal-phase elimination rate constant, slope of curves terminal segment at semi-log concentration-time curve calculated by linear regression.
AUC_%Extrap | Up to 72 hours post-dose of each drug
  The percentage of the AUC0-inf that has been extrapolated. AUC_%Extrap = [(AUC0-∞-AUC0-t)/AUC0-∞] × 100%
CL/F | Up to 72 hours post-dose of each drug
  Total body clearance after single dose. CL/F = Dose/AUC0-inf
Vz/F | Up to 72 hours post-dose of each drug
  apparent volume of distribution after single dose. Vz/F = Dose/AUC0-∞/λz
MRT0-t | Up to 72 hours post-dose of each drug
  Mean residence time within the time from time zero to the lowest testing plasma concentration after single dose. MRT0-t = AUMC0-t/AUC0-t
MRT0-∞ | Up to 72 hours post-dose of each drug
  Mean residence time extrapolated from zero to infinity after single dose. MRT 0-∞ = AUMC 0-∞/AUC 0-∞.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Tiantan Hospital, Capital Medical University Beijing, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No